CLINICAL TRIAL: NCT02921256
Title: A Phase II Clinical Trial Platform of Sensitization Utilizing Total Neoadjuvant Therapy (TNT) in Rectal Cancer
Brief Title: Veliparib, Pembrolizumab, and Combination Chemotherapy in Treating Patient With Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-00222; NCI-2016-00222 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GI002; s17-00197; NRG-GI002 (Other: NRG Oncology); NRG-GI002 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2016-09-30; First posted 2016-10-03 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Rectal Adenocarcinoma; Stage II Rectal Cancer AJCC v7; Stage III Rectal Cancer AJCC v7
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Fluorouracil; dehydroftorafur; Radiotherapy, Intensity-Modulated; Leucovorin; Oxaliplatin; pembrolizumab; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (mFOLFOX6, RT, capecitabine) (Active Comparator): Patients receive mFOLFOX6 regimen consisting of oxaliplatin IV over 2 hours on day 1, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last does of mFOLFOX6 patient undergo RT and receive capecitabine PO BID Monday-Friday for 5 weeks in the absence of disease progression or unacceptable toxicity. Participants assigned to Arm I concurrently with Arm II or with Arm III.
  Interventions: Drug: Capecitabine; Drug: Fluorouracil; Radiation: Intensity-Modulated Radiation Therapy; Drug: Leucovorin; Drug: Oxaliplatin
- Arm II (mFOLFOX6, RT, capecitabine, veliparib) (Experimental): Patients receive mFOLFOX6 regimen consisting of oxaliplatin IV over 2 hours on day 1, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for up to 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last does of mFOLFOX6 patient undergo RT and receive capecitabine PO BID and veliparib PO BID Monday-Friday for 5 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Fluorouracil; Radiation: Intensity-Modulated Radiation Therapy; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Veliparib
- Arm III (mFOLFOX6, RT, capecitabine, pembrolizumab) (Experimental): ARM III: Patients receive mFOLFOX6 regimen consisting of oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last does of mFOLFOX6 patient undergo RT and receive capecitabine PO BID Monday-Friday for 5 weeks. They also receive pembrolizumab IV over 30 minutes every 3 weeks beginning on day 1 of RT for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Fluorouracil; Radiation: Intensity-Modulated Radiation Therapy; Drug: Leucovorin; Drug: Oxaliplatin; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Radiation: Intensity-Modulated Radiation Therapy — Undergo intensity modulated radiation therapy
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; Keytruda; Lambrolizumab; MK-3475; Pembrolizumab Biosimilar BCD-201; SCH 900475
  Arms: Arm III (mFOLFOX6, RT, capecitabine, pembrolizumab)
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888
  Arms: Arm II (mFOLFOX6, RT, capecitabine, veliparib)

SUMMARY:
This randomized phase II trial studies how well veliparib or pembrolizumab work with combination chemotherapy and radiation therapy in treating patients with rectal cancer that has spread from where it started to nearby tissue or lymph nodes (locally advanced). Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as modified (m)FOLFOX6 regimen, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving veliparib or pembrolizumab with combination chemotherapy and radiation therapy may kill more tumor cells, make the tumor smaller, and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate an absolute improvement in neoadjuvant rectal cancer (NAR) score for the experimental regimen as compared to concurrently randomized control patients.

SECONDARY OBJECTIVES:

I. To compare overall survival (OS). II. To compare disease-free survival (DFS). III. To compare the rate of pathologic complete response (pCR) (nodes and tumor).

IV. To compare the rate of sphincter preservation.

TERTIARY OBJECTIVES:

I. To compare the proportion of patients who have a tumor resection overall, conditional on beginning induction chemotherapy, and conditional on beginning chemoradiotherapy.

II. To compare time from initiation of chemoradiotherapy to surgery in the subset of patients with tumor resection.

EXPLORATORY OBJECTIVES:

I. To estimate the rate of disease progression during chemotherapy (prior to chemoradiation).

II. To compare the rate of clinical complete response rate (cCR). III. To compare the rate of negative circumferential margin. IV. To compare the rate of completion of all cycles of neoadjuvant chemotherapy.

V. To compare the rate of completion of full course of chemoradiation. VI. To compare the toxicity and safety between interventions. VII. To explore the correlative molecular predictors of response and distant failure.

VIII. To explore the relationship between radiographic findings and pathologic outcomes.

OUTLINE: Patients are sequentially randomized to treatment arms, initially ARM I or ARM II and then later either ARM I or ARM III.

ARM I: Patients receive mFOLFOX6 regimen consisting of oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last does of mFOLFOX6 patient undergo radiation therapy (RT) and receive capecitabine orally (PO) twice daily (BID) Monday-Friday for 5 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive mFOLFOX6 regimen consisting of oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last does of mFOLFOX6 patient undergo RT and receive capecitabine PO BID and veliparib PO BID Monday-Friday for 5 weeks in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive mFOLFOX6 regimen consisting of oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last does of mFOLFOX6 patient undergo RT and receive capecitabine PO BID Monday-Friday for 5 weeks. They also receive pembrolizumab IV over 30 minutes every 3 weeks beginning on day 1 of RT for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have signed and dated an Institutional Review Board (IRB)-approved consent form that conforms to federal and institutional guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Diagnosis of adenocarcinoma of the rectum with the major portion of the tumor intact; Note: prior to randomization, the investigator must specify and document each of the following:

  * Distance of the lowest tumor margin from the anal verge; and
  * Intent for sphincter sparing or non-sphincter sparing surgical resection according to the primary surgeon; and
  * The majority of the untreated tumor must be < 12 cm from the anal verge or below the peritoneal reflection as determined by the treating surgeon
* The tumor must be clinically determined to be locally advanced stage II or stage III rectal cancer, and must also meet any ONE of the following criteria:

  * Distal location (as defined by measurement on magnetic resonance imaging [MRI], transrectal ultrasound [ERUS]/pelvic computed tomography [CT] [with IV contrast] scan or palpable on digital rectal examination [DRE]): cT3-4 =< 5 cm from the anal verge, any N
  * Bulky: any cT4 or evidence that the tumor is adjacent to (defined as within 3 mm of) the mesorectal fascia on MRI or ERUS/pelvic CT (with IV contrast) scan
  * High risk for metastatic disease with 4 or more regional lymph nodes (cN2); clinical nodal or "cN" status for eligibility includes the total number of nodes (N2 = 4 or more) in the mesorectal and superior rectal stations measuring >= 1.0 cm in any axis on cross sectional or endoscopic imaging; Note: nodes must measure 1.0 cm or greater to be considered positive for this eligibility requirement
  * Not a candidate for sphincter-sparing surgical resection prior to neoadjuvant therapy (as planned by the primary surgeon)

    * Note: clinical stage of the primary tumor and nodes may be determined locally by rectal endoscopic ultrasound or pelvic MRI (pelvic MRI is strongly preferred); CT scan with IV contrast is acceptable provided there is evidence of T4 and/or N2 disease
* Patients must have the ability to swallow and retain oral medication
* Absolute neutrophil count (ANC) must be >= 1200/mm^3 (within 28 days before randomization)
* Platelet count must be >= 100,000/mm^3 (within 28 days before randomization)
* Hemoglobin must be >= 10 g/dL (within 28 days before randomization)
* Total bilirubin must be =< ULN (upper limit of normal) for the lab unless the patient has a bilirubin elevation > ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin (within 28 days before randomization)
* Alkaline phosphatase must be =< 3 x ULN for the lab (within 28 days before randomization)
* Aspartate aminotransferase (AST) must be =< 3 x ULN for the lab (within 28 days before randomization);

  * Note: if alanine aminotransferase (ALT) is performed instead of AST (per institution's standard practice), the ALT value must be =< 3 x ULN; if both were performed, the AST must also be =< 3 x ULN; if AST and/or ALT is >= ULN but =< 3 x ULN, serologic testing for hepatitis B and C must be performed and results for viral infection must be negative
* Serum creatinine =< ULN for the lab and measured or calculated creatinine clearance > 60 mL/min (within 28 days before randomization)
* Serum potassium, magnesium, and calcium levels within 28 days before randomization must be within normal limits (WNL) for the lab
* International normalized ratio of prothrombin time (INR) within 28 days before randomization must be =< ULN for the lab; patients who are therapeutically treated with an agent such as warfarin may participate if they are on a stable dose and no underlying abnormality in coagulation parameters exists per medical history
* Patients with acquired immunodeficiency syndrome (AIDS-related illnesses) or known human immunodeficiency virus (HIV) disease must:

  * Have a cluster of differentiation (CD)4 count >= 200 cells/uL within 30 days before beginning study therapy
  * Be off all antiretroviral therapy (prophylaxis/treatment) more than 60 days before beginning study therapy, and
  * Have no evidence of opportunistic infections
* Pregnancy test (urine or serum beta-human chorionic gonadotropin [HCG]) done within 72 hours before randomization must be negative (for women of childbearing potential only); if urine pregnancy results are positive or cannot be confirmed as negative, a serum pregnancy test will be required

Exclusion Criteria:

* Rectal cancer histology other than adenocarcinoma (i.e., sarcoma, lymphoma, squamous cell carcinoma, mucosal melanoma, etc.)
* Definitive clinical or radiologic evidence of metastatic disease; required imaging studies must have been performed within 28 days prior to randomization; Note: Distant clinical staging to exclude patients with overt metastatic disease is determined by:

  * Chest: CT scan (preferred); chest x-ray posterioranterior (PA) and lateral (acceptable); or positron emission tomography (PET) scan (acceptable)
  * Abdomen: CT scan with IV contrast (preferred); or MRI (acceptable)
  * Pelvis: MRI (preferred) or CT scan with IV contrast (acceptable)

    * (It is recommended that the same imaging tests that are performed before randomization be used at follow-up time points; Note: CT scans of the abdomen and pelvis must be performed with IV contrast)
* History of prior invasive rectal malignancy, regardless of disease-free interval
* Cardiac disease that would preclude the use of any of the drugs included in the GI002 treatment regimen; this includes but is not limited to:

  * Clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or indwelling temporary pacemaker
  * Ventricular tachycardia or supraventricular tachycardia that requires treatment with class Ia antiarrhythmic drugs (e.g., quinidine, procainamide, disopyramide) or class III antiarrhythmic drug (e.g., sotalol, amiodarone, dofetilide); use of other antiarrhythmic drugs is permitted
  * Second- or third-degree atrioventricular (AV) block unless treated with a permanent pacemaker
  * Complete left bundle branch block (LBBB)
  * History of long QT syndrome
  * Corrected QT (QTc) >= 450 ms
* Sensory or motor neuropathy >= grade 2
* History of, or any evidence of active, non-infectious pneumonitis
* Active inflammatory bowel disease (i.e., patients requiring current medical interventions or who are symptomatic) or have a history of abdominal surgery or other medical condition that may, in the opinion of the treating physician, interfere with gastrointestinal motility or absorption
* Active autoimmune disease that has required systemic treatment within the past 2 years (i.e., with use of modifying agents, corticosteroids, or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* History of active TB (Bacillus tuberculosis)
* Active or chronic infection requiring systemic therapy
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study therapy; the use of physiologic doses of corticosteroids may be approved after consultation with the study principal investigator (PI)
* Active seizure disorder uncontrolled by medication
* Any antineoplastic therapy for this cancer before randomization
* Synchronous colon cancer
* Other invasive cancer within 5 years before randomization; exceptions are colonic polyps, non-melanoma skin cancer or carcinoma-in-situ of the cervix
* Antineoplastic therapy (e.g. chemotherapy or targeted therapy) for other invasive cancer within 5 years before randomization; (for the purposes of this study, hormonal therapy is not considered chemotherapy)
* Prior treatment with an investigational compound being tested in this study (e.g., poly ADP ribose polymerase [PARP] inhibitor, anti-PD-1, anti-PD-L1, or anti-PD-L2)
* Receipt of live vaccination within 28 days before randomization; seasonal flu vaccines that do not contain live virus are permitted
* Major surgery within 4 weeks before randomization
* Any therapeutic pelvic radiation
* Known homozygous DPD (dihydro pyrimidine dehydrogenase) deficiency
* Any of the following because this study involves agents that have known or potential genotoxic or mutagenic, and teratogenic effects:

  * Pregnant women
  * Nursing women who are unwilling to discontinue nursing
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (e.g., hormonal or barrier method of birth control; abstinence) for the duration of study treatment and for 4 months after the last dose of study therapy
* Co-morbid illnesses or other concurrent disease that, in the judgement of the clinician obtaining informed consent, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens or prevent required follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J George, Principal Investigator — NRG Oncology
Locations (650):
- United States (645):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Southern Cancer Center PC-Mobile, Mobile, Alabama
  - Southern Cancer Center PC-Providence, Mobile, Alabama
  - Southern Cancer Center PC-Springhill, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Enloe Medical Center, Chico, California
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - William Backus Hospital, Norwich, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Genesis Cancer Center - Silvis, Silvis, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center - 68th Street Place, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Garnet Health Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - The West Clinic - Wolf River, Germantown, Tennessee
  - The West Clinic - Mid-Town, Memphis, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Leigh Hospital, Norfolk, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Tri-Cities Cancer Center, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - FHCC South Lake Union, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Puerto Rico (5):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Hall WA, Li J, You YN, Gollub MJ, Grajo JR, Rosen M, dePrisco G, Yothers G, Dorth JA, Rahma OE, Russell MM, Gross HM, Jacobs SA, Faller BA, George S, Al Baghdadi T, Haddock MG, Valicenti R, Hong TS, George TJ. Prospective Correlation of Magnetic Resonance Tumor Regression Grade With Pathologic Outcomes in Total Neoadjuvant Therapy for Rectal Adenocarcinoma. J Clin Oncol. 2023 Oct 10;41(29):4643-4651. doi: 10.1200/JCO.22.02525. Epub 2023 Jul 21. PMID 37478389
- [Derived] Rahma OE, Yothers G, Hong TS, Russell MM, You YN, Parker W, Jacobs SA, Colangelo LH, Lucas PC, Gollub MJ, Hall WA, Kachnic LA, Vijayvergia N, O'Rourke MA, Faller BA, Valicenti RK, Schefter TE, George S, Kainthla R, Stella PJ, Sigurdson E, Wolmark N, George TJ. Use of Total Neoadjuvant Therapy for Locally Advanced Rectal Cancer: Initial Results From the Pembrolizumab Arm of a Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 Aug 1;7(8):1225-1230. doi: 10.1001/jamaoncol.2021.1683. PMID 34196693

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (mFOLFOX6, RT, Capecitabine): Patients receive mFOLFOX6 regimen consisting of oxaliplatin IV over 2 hours on day 1, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last does of mFOLFOX6 patient undergo RT and receive capecitabine PO BID Monday-Friday for 5 weeks in the absence of disease progression or unacceptable toxicity. Participants assigned to Arm I concurrently with Arm II are described as Arm Ia and participants assigned to Arm I concurrently with Arm III are described as Arm Ib.
  Capecitabine: Given PO
  Fluorouracil: Given IV
  Intensity-Modulated Radiation Therapy: Undergo intensity modulated radiation therapy
  Leucovorin: Given IV
  Oxaliplatin: Given IV
Period: Arm 1a v. Arm II
Arm/Group | Arm I (mFOLFOX6, RT, Capecitabine) | Arm II (mFOLFOX6, RT, Capecitabine, Veliparib) | Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab)
Started | 88 | 90 | 0
Completed | 72 | 57 | 0
Not Completed | 16 | 33 | 0
Not completed — Adverse Event | 6 | 15 | 0
Not completed — Death | 0 | 2 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 9 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 6 | 0
Period: Arm Ib v Arm III
Arm/Group | Arm I (mFOLFOX6, RT, Capecitabine) | Arm II (mFOLFOX6, RT, Capecitabine, Veliparib) | Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab)
Started | 95 | 0 | 90
Completed | 71 | 0 | 75
Not Completed | 24 | 0 | 15
Not completed — Adverse Event | 9 | 0 | 4
Not completed — Death | 1 | 0 | 1
Not completed — Lack of Efficacy | 2 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 3
Not completed — Physician Decision | 4 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm Ia (mFOLFOX6, RT, Capecitabine): Participants assigned to active comparator arm concurrent to Arm II.Patients receive mFOLFOX6 regimen consisting of oxaliplatin IV over 2 hours on day 1, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last does of mFOLFOX6 patient undergo RT and receive capecitabine PO BID Monday-Friday for 5 weeks in the absence of disease progression or unacceptable toxicity.
  Capecitabine: Given PO
  Fluorouracil: Given IV
  Intensity-Modulated Radiation Therapy: Undergo intensity modulated radiation therapy
  Leucovorin: Given IV
  Oxaliplatin: Given IV
- Arm Ib (mFOLFOX6, RT, Capecitabine): Participants assigned to active comparator arm concurrent to Arm III. Patients receive mFOLFOX6 regimen consisting of oxaliplatin IV over 2 hours on day 1, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last does of mFOLFOX6 patient undergo RT and receive capecitabine PO BID Monday-Friday for 5 weeks in the absence of disease progression or unacceptable toxicity.
  Capecitabine: Given PO
  Fluorouracil: Given IV
  Intensity-Modulated Radiation Therapy: Undergo intensity modulated radiation therapy
  Leucovorin: Given IV
  Oxaliplatin: Given IV
- Total: Total of all reporting groups
Arm/Group | Arm Ia (mFOLFOX6, RT, Capecitabine) | Arm II (mFOLFOX6, RT, Capecitabine, Veliparib) | Arm Ib (mFOLFOX6, RT, Capecitabine) | Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab) | Total
Number analyzed (Participants) | 88 | 90 | 95 | 90 | 363
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (10.9) | 56.0 (9.8) | 55.7 (11.2) | 55.5 (11.1) | 55.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 29 | 30 | 117
  Male | 59 | 61 | 66 | 60 | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 5 | 9 | 18
  Not Hispanic or Latino | 84 | 86 | 83 | 78 | 331
  Unknown or Not Reported | 1 | 3 | 7 | 3 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 1 | 4
  Asian | 2 | 8 | 4 | 3 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 4 | 7 | 6 | 2 | 19
  White | 76 | 71 | 77 | 77 | 301
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 5 | 3 | 6 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Neoadjuvant Rectal Cancer (NAR) Score
Description: A linear regression model that controls for the stratification factors (cT-stage and cN-stage) will be used. Mean NAR scores along with standard errors and confidence intervals will be reported by treatment. The NAR score ranges from zero to 100 with lower values corresponding to better prognosis.
Time Frame: Baseline to up to 3 years
Population: Patients who had a tumor resection and have pathology o the tumor specimen were evaluable for the primary endpoint of NAR score and included in the analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Arm Ia (mFOLFOX6, RT, Capecitabine): Participants assigned to active comparator arm concurrent to Arm II. Patients receive mFOLFOX6 regimen consisting of oxaliplatin IV over 2 hours on day 1, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last does of mFOLFOX6 patient undergo RT and receive capecitabine PO BID Monday-Friday for 5 weeks in the absence of disease progression or unacceptable toxicity.
  Capecitabine: Given PO
  Fluorouracil: Given IV
  Intensity-Modulated Radiation Therapy: Undergo intensity modulated radiation therapy
  Leucovorin: Given IV
  Oxaliplatin: Given IV
- Arm Ib (mFOLFOX6, RT, Capecitabine): Participants assigned to active comparator arm concurrent to ARM III. Patients receive mFOLFOX6 regimen consisting of oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last does of mFOLFOX6 patient undergo RT and receive capecitabine PO BID Monday-Friday for 5 weeks in the absence of disease progression or unacceptable toxicity.
  Capecitabine: Given PO
  Fluorouracil: Given IV
  Intensity-Modulated Radiation Therapy: Undergo intensity modulated radiation therapy
  Leucovorin: Given IV
- Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab): ARM III: Patients receive mFOLFOX6 regimen consisting of oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. 3-4 weeks after last dose of mFOLFOX6 patient undergoes RT and receives capecitabine PO BID Monday-Friday for 5 weeks. They also receive pembrolizumab IV over 30 minutes every 3 weeks beginning on day 1 of RT for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Capecitabine: Given PO
  Fluorouracil: Given IV
  Intensity-Modulated Radiation Therapy: Undergo intensity modulated radiation therapy
  Leucovorin: Given IV
  Oxaliplatin: Given IV
  Pembrolizumab:Given IV
Arm/Group | Arm Ia (mFOLFOX6, RT, Capecitabine) | Arm II (mFOLFOX6, RT, Capecitabine, Veliparib) | Arm Ib (mFOLFOX6, RT, Capecitabine) | Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab)
Number analyzed (Participants) | 72 | 68 | 68 | 69
score on a scale | 12.6 [9.8 to 15.3] | 13.7 [10.2 to 17.2] | 14.1 [10.7 to 17.4] | 11.5 [8.5 to 14.5]
Statistical Analysis 1: Comparison: Arm Ia (mFOLFOX6, RT, Capecitabine) vs Arm II (mFOLFOX6, RT, Capecitabine, Veliparib); Test type: Superiority; p = 0.69, Regression, Linear
Statistical Analysis 2: Comparison: Arm Ib (mFOLFOX6, RT, Capecitabine) vs Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab); Test type: Superiority; p = 0.26, Regression, Linear

2. Secondary Outcome: Overall Survival
Description: Analyzed using the stratified log rank test with strata cT-stage and cN-stage. Kaplan-Meier plots will illustrate the distribution of these endpoints by treatment. Cox regression models will be used to estimate hazard ratios and associated confidence intervals.
Time Frame: Time from randomization, assessed up to 3 years
Population: Participants with follow-up
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm Ia (mFOLFOX6, RT, Capecitabine) | Arm II (mFOLFOX6, RT, Capecitabine, Veliparib) | Arm Ib (mFOLFOX6, RT, Capecitabine) | Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab)
Number analyzed (Participants) | 86 | 89 | 90 | 85
proportion of participants | 0.922 [0.834 to 0.964] | 0.849 [0.754 to 0.910] | 0.867 [0.772 to 0.924] | 0.950 [0.870 to 0.981]

3. Secondary Outcome: Disease Free Survival
Description: as for outcome 2
Time Frame: Time from randomization, assessed up to 3 years
Population: Participants with follow-up
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm Ia (mFOLFOX6, RT, Capecitabine) | Arm II (mFOLFOX6, RT, Capecitabine, Veliparib) | Arm Ib (mFOLFOX6, RT, Capecitabine) | Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab)
Number analyzed (Participants) | 86 | 89 | 90 | 85
proportion of participants | 0.675 [0.559 to 0.766] | 0.600 [0.490 to 0.694] | 0.638 [0.528 to 0.729] | 0.636 [0.522 to 0.730]

4. Secondary Outcome: Rate of Pathologic Complete Response (Nodes and Tumor) ypT0 and ypN0
Description: Pathologic Complete Response means no remaining cancer detectable in the pathology sample. Analyzed by a logistic regression model that controls for the stratification factors (cT-stage and cN-stage). Observed proportions along with confidence intervals will be presented by treatment.
Time Frame: Up to 3 years
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm Ia (mFOLFOX6, RT, Capecitabine) | Arm II (mFOLFOX6, RT, Capecitabine, Veliparib) | Arm Ib (mFOLFOX6, RT, Capecitabine) | Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab)
Number analyzed (Participants) | 74 | 71 | 68 | 69
percentage of participants | 21.6 [12.9 to 32.7] | 33.8 [23.0 to 46.0] | 29.4 [19.0 to 41.7] | 31.9 [21.2 to 44.2]

5. Secondary Outcome: Rate of Sphincter Preservation
Description: Sphincter preservation means that the surgical procedure used to remove the tumor did not disturb the sphincter muscle. Analyzed by a logistic regression model that controls for the stratification factors (cT-stage and cN-stage). Observed proportions along with confidence intervals will be presented by treatment.
Time Frame: Up to 3 years
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm Ia (mFOLFOX6, RT, Capecitabine): Arm Ia (mFOLFOX6, RT, capecitabine)
- Arm II (mFOLFOX6, RT, Capecitabine, Veliparib): Arm II (mFOLFOX6, RT, capecitabine, veliparib)
- Arm Ib (mFOLFOX6, RT, Capecitabine, Pembrolizumab): Arm Ib (mFOLFOX6, RT, capecitabine)
- Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab): Arm III (mFOLFOX6, RT, capecitabine, pembrolizumab)
Arm/Group | Arm Ia (mFOLFOX6, RT, Capecitabine) | Arm II (mFOLFOX6, RT, Capecitabine, Veliparib) | Arm Ib (mFOLFOX6, RT, Capecitabine, Pembrolizumab) | Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab)
Number analyzed (Participants) | 80 | 81 | 69 | 69
percentage of participants | 52.5 [41.0 to 63.8] | 59.3 [47.8 to 70.1] | 71.0 [58.8 to 81.3] | 59.4 [46.9 to 71.1]

6. Other Pre Specified Outcome: Proportion of Patients Who Have a Tumor Resection Overall (and Conditional on Beginning Induction Chemotherapy, and Conditional on Beginning Chemoradiotherapy)
Description: Analyzed by a logistic regression model that controls for the stratification factors (cT-stage and cN-stage). Observed proportions along with confidence intervals will be presented by treatment.
Time Frame: Up to 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Time From Initiation of Chemoradiotherapy to Surgery in the Subset of Patients With Tumor Resection
Description: Analyzed using the stratified log rank test with strata cT-stage and cN-stage. Kaplan-Meier plots will illustrate the distribution of time to surgery (TTS) by treatment. Cox regression models will be used to estimate hazard ratios and associated confidence intervals.
Time Frame: Up to 3 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Rate of Disease Progression During Chemotherapy (Prior to Chemoradiation)
Description: as for outcome 6
Time Frame: Up to 3 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Rate of Clinical Complete Response Rate, ycT0
Description: as for outcome 6
Time Frame: Up to 3 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Rate of Negative Circumferential Margin
Description: as for outcome 6
Time Frame: Up to 3 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Rate of Completion of All Cycles of Neoadjuvant Chemotherapy
Description: as for outcome 6
Time Frame: Up to 3 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Rate of Completion of Full Course of Chemoradiation
Description: as for outcome 6
Time Frame: Up to 3 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Incidence of Toxicity Including Patient-reported Toxicities
Description: Will be assessed using Common Terminology for Adverse Events (CTCAE) version 4.0 (CTCAE version 5.0 beginning April 1, 2018).
Time Frame: 30 days after last study treatment
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Correlative Molecular Predictors of Response and Distant Failure
Description: Cox regression models will be used to evaluate markers for time-to-event variables. Logistic regression models will be used for binary variables. Models will control for stratification factors and possibly other prognostic variables (e.g. gender or treatment).
Time Frame: Up to 3 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Relationship Between Radiographic Findings and Pathologic Outcomes
Description: Will explore the relationship between radiographic findings and pathologic outcomes.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Deaths were assessed for up to 3 years. Adverse Events were assessed from study entry to surgery, about 7 months.
Description: Participants at Risk includes any patient who submitted an AE form. Not all participants returned Adverse Event forms; therefore, the Number of Participants At Risk differs between All-Cause Mortality and Serious/Other Adverse Events.
Groups:
- Arm Ib (mFOLFOX6, RT, Capecitabine): Arm Ib (mFOLFOX6, RT, capecitabine)
- Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab): Arm Ib (mFOLFOX6, RT, capecitabine, pembrolizumab)
Arm/Group | Arm Ia (mFOLFOX6, RT, Capecitabine) | Arm II (mFOLFOX6, RT, Capecitabine, Veliparib) | Arm Ib (mFOLFOX6, RT, Capecitabine) | Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 7/87 | 14/90 | 13/93 | 6/87
Serious Adverse Events (participants affected / at risk) | 16/83 | 25/88 | 21/84 | 15/82
Other Adverse Events (participants affected / at risk) | 83/83 | 86/88 | 82/84 | 81/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm Ia (mFOLFOX6, RT, Capecitabine) (N=83) | Arm II (mFOLFOX6, RT, Capecitabine, Veliparib) (N=88) | Arm Ib (mFOLFOX6, RT, Capecitabine) (N=84) | Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab) (N=82)
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Anaphylaxis (Immune system disorders) | 1 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 3 | 1 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 1 | 0
Delusions (Psychiatric disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 7 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Fever (General disorders) | 0 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 6 | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rectal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Renal calculi (Renal and urinary disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0
Thromboembolic event (Vascular disorders) | 3 | 1 | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Pelvic infection (Infections and infestations) | 0 | 1 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 2 | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 4 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 1 | 1 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rectal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestine infection (Infections and infestations) | 0 | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rectal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm Ia (mFOLFOX6, RT, Capecitabine) (N=83) | Arm II (mFOLFOX6, RT, Capecitabine, Veliparib) (N=88) | Arm Ib (mFOLFOX6, RT, Capecitabine) (N=84) | Arm III (mFOLFOX6, RT, Capecitabine, Pembrolizumab) (N=82)
Abdominal pain (Gastrointestinal disorders) | 10 | 21 | 7 | 6
Alanine aminotransferase increased (Investigations) | 2 | 5 | 10 | 8
Anal pain (Gastrointestinal disorders) | 12 | 19 | 2 | 6
Anemia (Blood and lymphatic system disorders) | 11 | 18 | 13 | 14
Anorexia (Metabolism and nutrition disorders) | 12 | 24 | 15 | 4
Anxiety (Psychiatric disorders) | 3 | 8 | 6 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 7 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 5 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 7 | 0
Constipation (Gastrointestinal disorders) | 13 | 13 | 13 | 10
Dehydration (Metabolism and nutrition disorders) | 9 | 21 | 12 | 5
Depression (Psychiatric disorders) | 2 | 5 | 1 | 4
Diarrhea (Gastrointestinal disorders) | 30 | 43 | 29 | 25
Dysgeusia (Nervous system disorders) | 3 | 7 | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 8 | 3
Fatigue (General disorders) | 26 | 46 | 33 | 32
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 | 5 | 0 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 8 | 5 | 2
Hypertension (Vascular disorders) | 24 | 16 | 19 | 24
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 6 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 8 | 6 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 5 | 4 | 3
Hypokalemia (Metabolism and nutrition disorders) | 7 | 10 | 7 | 11
Hypotension (Vascular disorders) | 7 | 5 | 1 | 3
Hypothyroidism (Endocrine disorders) | 0 | 0 | 9 | 1
Infections and infestations - Other, specify (Infections and infestations) | 3 | 1 | 5 | 4
Insomnia (Psychiatric disorders) | 5 | 3 | 5 | 3
Lymphocyte count decreased (Investigations) | 35 | 37 | 36 | 25
Mucositis oral (Gastrointestinal disorders) | 10 | 11 | 4 | 7
Nausea (Gastrointestinal disorders) | 21 | 34 | 24 | 19
Neutrophil count decreased (Investigations) | 36 | 50 | 40 | 34
Pain (General disorders) | 5 | 2 | 6 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 5
Paresthesia (Nervous system disorders) | 3 | 8 | 6 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 5 | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 18 | 21 | 25 | 26
Platelet count decreased (Investigations) | 10 | 15 | 21 | 15
Proctitis (Gastrointestinal disorders) | 6 | 8 | 6 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3 | 5 | 3
Rectal pain (Gastrointestinal disorders) | 7 | 13 | 16 | 12
Thromboembolic event (Vascular disorders) | 10 | 4 | 7 | 6
Urinary tract infection (Infections and infestations) | 3 | 5 | 7 | 6
Vomiting (Gastrointestinal disorders) | 8 | 14 | 13 | 3
Weight loss (Investigations) | 3 | 11 | 6 | 5
White blood cell decreased (Investigations) | 11 | 28 | 22 | 23
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 3 | 10 | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 4 | 4 | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 14 | 18 | 12 | 13
Rectal mucositis (Gastrointestinal disorders) | 4 | 8 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 3 | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT02921256/Prot_SAP_000.pdf